CLINICAL TRIAL: NCT00277407
Title: An Investigation Into the Outcome of NAET Treatment on Children With Allergy-Related Autism Spectrum Disorders in a Multi-Clinical Setting.
Brief Title: Treatment of Autistic Children Using NAET Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nambudripad's Allergy Research Foundation (Other)
Collaborators: Anonymous (Ambiguous)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MulticlinicalAutism Study; NARFoundationAutismStudy2006
Record Dates: First submitted 2006-01-12; First posted 2006-01-16 (Estimated); Last update posted 2007-05-07 (Estimated); Status verified 2007-05

CONDITIONS: Autism; Food Allergies
Keywords: NAET; Chiropractic procedures; Acupuncture/acupressure; Treatment of Autism by holistic procedures; Food and Vaccination allergy
MeSH Terms: conditions — Autistic Disorder; Food Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: NAET with acupressure and/or chiropractic procedures

SUMMARY:
1. Purpose of this study is to determine whether NAET procedures are effective in the treatment of children with allergy-related autism spectrum disorders in restoring their verbal and nonverbal communication.
2. Hypothesis: Children in the experimental group will show a significant improvement over the control group in verbal and nonverbal communication as most food allergen groups, environmental allergen groups, childhood immunizations, and some other relevant allergenic substances are desensitized in a systematic way using NAET® procedures within the specified period of study.

DETAILED DESCRIPTION:
A multi-clinical study on Children with Autism spectrum disorders Using NAET Nambudripad's Allergy Elimination Techniques) Treatments.

Participating NAET CLINIC LOCATIONS IN THE COUNTRY:

1. Mala Moosad, R.N., L.Ac., N.D. (Acupuncture, Allergies, NAET) Clinical Director, PNIB Research Center, 6714-36 Beach Blvd., Buena Park, CA 90621 Phone: (714) 523- 2817; Fax: (714) 523-3068. email: pnibquestions@yahoo.com
2. Robert Prince, M.D. (Psychiatry, NAET) and Iris Prince, R.N. NAET of North Carolina 1955 Woodberry Road, Charlotte, NC 28218. Phone: (704) 537-0221. E. mail: RMPrince@bellsouth.net
3. Ross Stark, BSEE, D. Ac., L.Ac 1925 Sleepy Hollow Lane, Annapolis, MD 21401 USA Phone: 410 266 3350. starktcm@starktcm.com
4. James Benjamin, M.D., and Joyce Benjamin, R.N. 7507 Old Chapel Dr. Bowie, MD 20715 USA Phone: 301 805 8399 Fax: 301 805 9417. E. mail: jj1987@verizon.net
5. Anthony De Siena, D.C. (Chiropractic, NAET, Allergies). Washington Street Chiropractic Center, LLC 771 Washington Street, Eugene, OR 97401 USA Phone: (541) 686-2225 Fax: 541 687 6975. E. mail: adesiena@juno.com
6. Nancy B. Rosen, R.N., M.Ac., L.Ac. 114 Lowell Ave Newtonville, MA 02460-1503 USA Phone: 617 558 7619 E.mail: NBR001@aol.com
7. Mira A. Champaneria, BDS 67 Lakewood Ave, Clear Grove, NJ 07009. Phone. (973) 699-1013. fax.(973) 239-5425 E. mail: mirachamp@hotmail.com
8. Sue Anderson, D.C.(Chiropractic, NAET). 2160 Huron Pkwy, Suite 1 Ann Arbor, MI 48104 USA Phone: (734) 973-9692. E. mail: sue.anderson@worldnet.att.net
9. Ray Alexander, D.C. (Chiropractic and Acupuncture) Alexander Chiropractic Clinic, 911 Duluth Hwy. N.W. Ste. B6 Lawrenceville, GA 30043 USA Phone: 770 339 1311 Fax: 770 339 3608.E. mail: drrayalex@aol.com
10. Marilyn Chernoff, N.D., Ph.D. 1924 Juan Tabo, Suite A, Albuquerque, NM 87112 Phone: 505 292 2222 Fax: 505 292 2771. e. mail: dr.marilyn@earthlink.net
11. Marilyn Elliott, D.C. (Chiropractic and NAET) 226 Clairmont Rd, Sterrett, AL 35147 Phone. (205) 980-4498. e. mail: drelliott@greystonechiropractic.com
12. Kathleen Jackson, NMD, RPh 10406 Spencer Hwy (W. Main), Suite B La Porte, TX 77571 Phone: 281 470 7300 Fax: 281 470 1386. e. mail: patk13@pdq.net
13. Farangis Tavily, L.Ac.(Acupuncture, Allergies, NAET) 20 Sunnyside Ave. A397 Mill Valley, CA 94941 USA Phone: (415) 302-7907. E. mail: inthenameofgod@sbcglobal.net.
14. Murray Lawson, D.C., D.A.C.N.B. (Chiropractic and NAET) Yavapai Neurology Center, 3755 Karicio Lane, Suite 2-A Prescott, AZ 86303 E. mail: 928 708 9144 Fax: 928 708 9156, drmjl@cableone.net
15. Gary Erkfritz, D.C. (Chiropractic, Allergies, NAET) 187 East Wilbur, Suite 1 Thousand oaks, CA 91360 USA Phone: 805 371 8082. E. mail: geedc@adelphia.net
16. Roya Nikzad, L.Ac., Ph.D. (Acupuncture, NAET). 8950 Villa La Jolla Dr., Suite C-117 La Jolla (San Diego), CA 92037 USA Phone: (858) 202-0322.E. mail: nikzr@aol.com
17. Margaret Owen, B.S., M.ED., N.D. 4105 Medical Parkway #202 Austin, TX 78756 Phone: 512 206 4158. email: mowens3108@msn.com
18. Yvonne Tyson, M.D., (Family Medicine, Board Certified in Acupuncture, Board Certified in Holistic Medicine, NAET) Alternate phone: (562) 498-0606. fax: (562) 423-0396.E. mail: tysonmd99@hotmail.com
19. Dave nelson, Ph.D. (Nutrition & NAET) Center for Advanced Medicine 4403 Manchester Ave., #107, Encinitas, CA 92024 Phone: 760 632-9042, Fax:: 760 632- 0574. E. mail: dccnelson2000@cox.net
20. John Crandall, DC (Chiropractic and NAET) 247 west 35th street, New York, NY 10001 Ph. 203 254 8445. E mail; drcrandall@naetnyc.com
21. Kathy Ferrante, L.Ch, CNHP 4353 edgewater drive, Suite # 3, Orlando, FL Ph. 407-297-0772 e. mail: adlwellness@juno.com
22. Roger Barnes, Dc, CCN 448 E. Main Street, Suite A, Bozeman, MT 59715 Ph. 406 585-7800. E. Mail: rogerbdc@aol.com

According to NAET theory, autism is a nutritional deficiency disorder causing biological, neurological and developmental problems in children. The nutritional deficiency is caused by poor digestion, absorption, assimilation and utilization of essential nutrients due to allergies. NAET is the only treatment known so far that is able to eliminate allergies permanently allowing the sufferer to live a normal life once again. NAET is a blend of medical knowledge and non-invasive painless, holistic treatment procedures that is able to eliminate various levels of sensitivities and allergies permanently to the treated allergens. In the past 22 years of our clinical practice, we have not seen any adverse reactions with NAET, if it is applied properly by a trained NAET practitioner.

ELIGIBILITY:
Inclusion Criteria:

all subjects (control and treatment group) should demonstrate typical autistic symptoms before beginning NAET® treatments: made no eye contact, unable to communicate verbally or nonverbally. All subjects should bring in a proof of established diagnosis of autism spectrum disorder by a conventional physician.

-

Exclusion Criteria:

Any child that has a history of various complications of illness other than autism spectrum disorder would be disqualified. Any patient who has any of the following conditions will also be disqualified.

1. Previous surgeries, congenital deformities of heart, lung, liver, brain, kidney, etc.
2. Any type of cancer
3. Aids
4. Any physically debilitating disorders and diagnosed mental retardation, Down's syndrome, etc.
5. Children with the history of severe allergies or anaphylactic reactions will be exclued.

   -

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2006-06; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Improvement in verbal and norverbal communication | Twenty-four months from the starting date (approximately may 2008)

SECONDARY OUTCOMES:
Reduction of commonly seen autistic traits | Twenty-four months from starting dat (May 2008)

CONTACTS AND LOCATIONS:
Overall Officials: Devi S. Nambudripad, DCLAcPhD, Principal Investigator — NAR Foundation
Locations (1):
- NAET Pain Clinic, Buena Park, California, United States